CLINICAL TRIAL: NCT02665260
Title: Randomized Pilot Study Investigating the Safety and Efficacy of Topical Cantharidin for the Treatment of Molluscum Contagiosum
Brief Title: Safety and Efficacy Study of Topical Cantharidin for the Treatment of Molluscum Contagiosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Steven R Cohen, Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-01-004
Record Dates: First submitted 2015-12-31; First posted 2016-01-27 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum | interventions — Cantharidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cantharidin with occlusion (Active Comparator): Cantharidin 0.7% topical with occlusion
  Interventions: Drug: Cantharidin; Device: Gauze occlusion bandage
- Cantharidin without occlusion (Experimental): Cantharidin 0.7% topical without occlusion
  Interventions: Drug: Cantharidin
- Placebo with occlusion (Placebo Comparator): Placebo topical with occlusion
  Interventions: Drug: Placebo; Device: Gauze occlusion bandage
- Placebo without occlusion (Placebo Comparator): Placebo topical without occlusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cantharidin — cantharidin 0.7% topical liquid
  Other Names: 2,6-Dimethyl-4,10-dioxatricyclo-decane-3,5-dione
  Arms: Cantharidin with occlusion; Cantharidin without occlusion
Drug: Placebo — Placebo topical liquid
  Other Names: flexible collodion
  Arms: Placebo with occlusion; Placebo without occlusion
Device: Gauze occlusion bandage — Gauze occlusion bandage with adhesive tape
  Arms: Cantharidin with occlusion; Placebo with occlusion

SUMMARY:
The purpose of this study is to determine if cantharidin is a safe and effective treatment for molluscum contagiosum in kids

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled trial. Participants were recruited from the Pediatric Dermatology clinic at Montefiore Medical Center. One hundred eligible participants were randomly assigned to receive cantharidin 0.7% topical, cantharidin 0.7% topical with occlusion, placebo, or placebo with occlusion. Treatments were applied at weeks 0 and 3 (blinded phase). At week 6, all participants were treated with open-label, topical cantharidin 0.7% without occlusion every 3 weeks until all lesions resolved (open-label phase).

ELIGIBILITY:
Inclusion Criteria:

* 2-17years
* Healthy
* <50 molluscum contagiosum lesions

Exclusion Criteria:

* Immunosuppressed
* Oral corticosteroids
* Sexually active/pregnant

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2012-07; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 6 subjects met exclusion criteria for having greater than 50 molluscum contagiosum lesions at screening.
Groups:
- Cantharidin With Occlusion: Patients treated with cantharidin 0.7% topical with occlusion
- Cantharidin Without Occlusion: Patients treated with cantharidin 0.7% topical without occlusion
- Placebo With Occlusion: Patients treated with placebo and occlusion
- Placebo Without Occlusion: Patients treated with placebo without conclusion
Period: Overall Study
Arm/Group | Cantharidin With Occlusion | Cantharidin Without Occlusion | Placebo With Occlusion | Placebo Without Occlusion
Started | 24 | 23 | 25 | 22
Completed | 22 | 22 | 21 | 21
Not Completed | 2 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cantharidin: Patients treated with 0.7% topical cantharidin without occlusion
- Cantharidin With Occlusion: Patients treated with 0.7% topical cantharidin with occlusion
- Placebo: Patients treated with placebo without occlusion
- Placebo With Occlusion: Patients treated with placebo vehicle with occlusion
- Total: Total of all reporting groups
Arm/Group | Cantharidin | Cantharidin With Occlusion | Placebo | Placebo With Occlusion | Total
Number analyzed (Participants) | 23 | 24 | 22 | 25 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 24 | 22 | 25 | 94
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 10 | 15 | 52
  Male | 9 | 11 | 12 | 10 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 22 | 16 | 13 | 17 | 68
  African American | 1 | 3 | 3 | 5 | 12
  Caucasian | 0 | 4 | 3 | 1 | 8
  Asian | 0 | 1 | 3 | 1 | 5
  Jamaican | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieve Complete Clearance at 6 Weeks
Description: Assess number of subjects who achieve a lesion count of zero at 6 weeks (end of open-label phase)
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cantharidin With Occlusion | Cantharidin Without Occlusion | Placebo With Occlusion | Placebo Without Occlusion
Number analyzed (Participants) | 24 | 23 | 25 | 22
Participants
  Number of subjects achieving lesion clearance | 10 | 7 | 2 | 3
  Number of subjects not achieving lesion clearance | 14 | 16 | 23 | 19

2. Secondary Outcome: Number of Subjects Who Experienced an Adverse Event
Description: Number of subjects who experienced an adverse event as assessed by patient-reported outcomes questionnaire at each visit
Time Frame: 33 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cantharidin | Cantharidin With Occlusion | Placebo | Placebo With Occlusion
Number analyzed (Participants) | 23 | 24 | 22 | 25
Participants
  Number experiencing adverse event | 0 | 0 | 0 | 0
  Number not experiencing adverse event | 23 | 24 | 22 | 25

ADVERSE EVENTS:
Groups:
- Cantharidin: Subjects treated with topical cantharidin 0.7% without occlusion
- Cantharidin With Occlusion: Subjects treated with topical cantharidin 0.7% with occlusion
- Placebo: Subjects treated with placebo without occlusion
- Placebo With Occlusion: Subjects treated with placebo with occlusion
Arm/Group | Cantharidin | Cantharidin With Occlusion | Placebo | Placebo With Occlusion
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/22 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No